CLINICAL TRIAL: NCT05111405
Title: A Randomized Prospective Multicenter Study Comparing Suture Button Suspensionplasty (SBS) with Ligament Reconstruction and Tendon Interposition (LRTI)
Brief Title: Study Comparing SBS and LRTI for Treatment of CMC Arthritis
Acronym: SBSvsLRTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FHREB # 2021-112
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, prospective trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trapezial excision with or without soft tissue interposition and /or ligament reconstruction (Other): The participating surgeon will perform their usual version of a trapeziectomy and thumb metacarpal using either FCR tendon or abductor hallucis longs (APL) tendon. Tendon interposition will be left to the surgeon's discretion.
  Interventions: Procedure: CMC Arthroplasty
- Suture button suspension arthroplasty (SBS) (Other): Dorso-radial incision, capsulotomy between extensor pollicis brevis (EPB) and APL protecting the radial artery. A second incision is made on dorsum of hand between the 2nd and 3rd MCs. A cannulated drill with suture passer is passed from base of 1st MC to mid 2nd MC. The TightropeTM is passed from 1st to second MC with one button on the base of the 1st MC. Trapeziectomy is then performed using a cruciate osteotomy and rongeurs. The thumb is adducted against index MC to avoid excessive tightening and the suture is tied over a second button on the 2nd MC. Closure of capsule with Vicryl. Closure of skin with running Prolene suture.
  Interventions: Procedure: CMC Arthroplasty

INTERVENTIONS:
Procedure: CMC Arthroplasty — Surgical intervention to treat CMC arthritis

SUMMARY:
A multi-center, randomized control trial comparing the two standard of care surgical treatments for CMC arthritis ; trapezial excision with or without soft tissue interposition and /or ligament reconstruction (LRTI) versus the suture button suspension arthroplasty (SBS). Patient reported outcomes will be collected at 6 and 6 weeks, 3, 6, and 12 months.

DETAILED DESCRIPTION:
LRTI is a well established treatment of CMC arthritis with good results.However, comparable results have also been reported with SBS, with the latter procedure eliminating the need for flexor carpi radialis (FCR) harvest and interposition, resulting in potential shorter OR time and donor site morbidity. To date, there have been biomechanical studies comparing LRTI vs suture button suspension arthroplasty (SBS), and clinical studies comparing trapeziectomy alone vs SBS, but to the best of our knowledge, no random control studies comparing LRTI with SBS.The primary objective is to determine whether treatment with SBS results in improved overall pain relief compared to LRTI as measured by patient reported outcomes.Secondary outcome measures will be to determine if SBS results in shorter OR time and improved grip and pinch strength compared to LRTI, as well as have comparable return to work times and amount of radiographic shortening as shown on radiographs (metacarpal shortening has been felt to lead to decreased grip strength).

ELIGIBILITY:
Inclusion Criteria:

* Age fifty years or older
* Isolated carpometacarpal (trapeziometacarpal) osteoarthritis
* Failure to respond to non-operative management
* Willing and able to consent on their own behalf and follow the protocol and clinical visits as described
* Able to read and understand English or have interpreter available

Exclusion Criteria:

* Previous surgery for CMC arthritis
* Duration of symptoms for less than 6 months
* Greater than or equal to 30 degrees of ipsilateral metacarpophalangeal (MCP) hyperextension
* Scaphotrapeziotrapezoidal (stage 4 CMC) arthritis
* Other significant ipsilateral wrist or hand pathology
* A history of inflammatory arthropathy
* A requirement for concomitant surgery for another condition
* Any previous hand or wrist fracture
* Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, not mentally competent to give consent, intellectually challenged patients without adequate support, etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale- Pain | 12 Months
  Participants overall assessment of their pain at maximal key pinch loading on a 10 cm visual analogue scale
Disabilities of the Arm, Shoulder and Hand Questionnaire | 12 Months
  A 30 Item questionnaire that measures an individuals' ability to complete tasks, absorb forces and severity of symptoms. Lower scores will indicated better outcomes.Lower scores will indicate better outcomes.
Patient Related Wrist Evaluation Questionnaire | 12 Months
  A 15 item questionnaire to measure wrist pain and disability pain in activities of daily living

SECONDARY OUTCOMES:
Operative Time | Intraoperative
  Time as recorded from the surgeons start of the procedure until the surgeons stop.
Strength | 12 Months
  Transverse volar grip strength as measured by a dynamometer and key and lateral pinch strength measure by a pinch gauge
Range of Motion | 12 Months
  Thumb flexion will be measured from the top of the thumb (pulp) to the base of the 5th metacarpal (pinky finger). Retropulsion measured as the distance between the thumb and table when the dorsum of the hand is pressed against the table.
Work Productivity and Activity Impairment: Specific Health Problem Questionnaire | 12 Months
  A questionnaire pertaining to the effect of the participant's CMC arthritis on their ability to work and perform regular activities. Lower scores will indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - South Campus Research Unit for Bone and Soft Tissue, Calgary, Alberta
  - Fraser Orthopaedic Research Society, New Westminster, British Columbia

IPD SHARING:
Plan to Share IPD: No